CLINICAL TRIAL: NCT04375800
Title: A Phase 2 Clinical Study to Evaluate the Pharmacokinetics, Safety, and Efficacy of Doravirine and Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate in Participants With HIV-1, Who Are 4 Weeks to Less Than 12 Years of Age and Weigh Less Than 45 kg
Brief Title: Doravirine (DOR) in Human Immunodeficiency Virus (HIV)-Infected Children Ages 4 Weeks to <12 Years and <45 kg (MK-1439-066)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1439-066; MK-1439-066 (Other: MSD); 2019-003955-13 (EudraCT Number)
Record Dates: First submitted 2020-05-04; First posted 2020-05-05 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Human Immunodeficiency Virus (HIV) Infection
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — doravirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Doravirine + 2 NRTIs (Experimental): Participants receive DOR (3.2 mg to 100 mg based on weight) in combination with 2 NRTIs (based on local label) for 96 weeks.
  Interventions: Drug: Doravirine; Drug: 2 NRTIs

INTERVENTIONS:
Drug: Doravirine — DOR capsules (3.2 to 100 mg); sachets (3.2 to 100 mg); or tablets (100 mg) taken once or twice daily by mouth.
  Other Names: MK-1439
Drug: 2 NRTIs — Participants receive 2 NRTIs per local label by mouth for 96 weeks as background therapy.

SUMMARY:
This is a single-group, open-label, multi-site study in pediatric participants with human immunodeficiency virus type 1 (HIV-1) infection, aged 4 weeks to <12 years and weighing <45 kg, who are treatment-naive (TN) or have been virologically suppressed (VS) on stable combination antiretroviral therapy (cART) for ≥3 months with no history of treatment failure. The first primary objective is to evaluate the steady state pharmacokinetics (PK) of doravirine (DOR) [MK-1439] when given in combination with 2 nucleoside/nucleotide analog reverse transcriptase inhibitors (NRTIs) or as part of the fixed dose combination (FDC) of DOR/lamivudine (3TC)/tenofovir disproxil fumarate (TDF) in participants ≥6 to <12 years and weighing ≥14 to <45 kg. The second primary objective is to evaluate the safety and tolerability of DOR when given with 2 NRTIs or as part of the FDC of DOR/3TC/TDF, in participants ≥6 to 12 years and weighing ≥14 to <45 kg, through Week 24.

DETAILED DESCRIPTION:
Participants who complete the Week 96 visit will be eligible to enroll in an Extension Study in which they may continue to receive DOR until it is commercially available, or for up to an additional 224 weeks (whichever comes first).

ELIGIBILITY:
Inclusion Criteria:

* Has HIV-1 infection confirmed at screening
* Has treatment history defined as either TN or with documented viral suppression (HIV-1 RNA <50 copies/mL) for ≥3 months on combination antiretroviral therapy (cART)
* Body weight is >3 kg to <45 kg
* If female, is not pregnant or breastfeeding, and one of the following applies:
* is not a woman of childbearing potential (WOCBP)
* is a WOCBP using an acceptable form of contraception, or is abstinent
* if a WOCBP must have a negative pregnancy test (urine or serum) within 24 hours of the first dose of study intervention

Study Extension Inclusion Criteria:

* Has completed the Week 96 visit.
* Is considered, in the opinion of the investigator, to have derived benefit from treatment with DOR plus the 2 NRTIs selected by the investigator, or DOR/3TC/TDF, by Week 96 of the study
* Is considered, in the opinion of the investigator, to be a clinically appropriate candidate for additional treatment with DOR plus 2 NRTIs selected by the investigator.
* Understands the procedures in the study extension and has provided (or have the participant's legally acceptable representative, if applicable, provide) documented informed consent/assent to enter the study extension and continue treatment with DOR plus 2 NRTIs selected by the investigator until DOR is available commercially in countries participating in the study or for up to an additional 224 weeks (whichever comes first).

Exclusion Criteria:

* Has evidence of renal disease
* Demonstrates evidence of liver disease
* Has clinical or laboratory evidence of pancreatitis
* Has any history of malignancy
* Has presence of any active acquired immunodeficiency syndrome (AIDS)-defining Opportunistic Infection
* Has an active diagnosis of hepatitis, including hepatitis B co-infection
* Has current active tuberculosis and/or is being treated with a rifampicin-containing regimen
* Has a medical condition that precludes absorption or intake of oral pellets/granules
* Has a history or current evidence of any condition, therapy, laboratory abnormality, or other circumstance that might confound results of the study or interfere with participating for the entire duration of the study
* Is taking or is anticipated to require systemic immunosuppressive therapy, immune modulators, or other prohibited therapy
* Is currently participating in or has participated in an interventional clinical study with an investigational compound or device from 45 days prior to Day 1 through the treatment period
* Has a documented or known virologic resistance to DOR
* Has any history of viremia (HIV RNA >1000 copies/mL) after at least 3 months on a non-nucleoside reverse transcriptase inhibitor (NNRTI)-based regimen

Ages: 4 Weeks to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Estimated)
Dates: Start 2021-02-03 (Actual); Primary Completion 2028-03-04 (Estimated); Study Completion 2034-04-11 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration-time curve from 0 to 24 hours postdose (AUC0-24hr) of DOR with 2 NRTIs in plasma at steady-state | Predose and 1, 2, 4, 12, and 24 hours postdose on Day 42
  Plasma AUC0-24 hr of DOR with 2 NRTIs will be determined at steady-state.
Maximum concentration (Cmax) of DOR with 2 NRTIs in plasma at steady-state | Predose and 1, 2, 4, 12, and 24 hours postdose on Day 42
  Plasma Cmax of DOR with 2 NRTIs will be determined at steady-state.
Concentration at 24 hours (C24) of DOR with 2 NRTIs in plasma at steady-state | 24 hours postdose on Day 42
  Plasma C24 of DOR with 2 NRTIs will be determined at steady-state.
Time to maximum concentration (Tmax) of DOR with 2 NRTIs in plasma at steady-state | Predose and 1, 2, 4, 12, and 24 hours postdose on Day 42
  Plasma Tmax of DOR with 2 NRTIs will be determined at steady-state.
Percentage of participants with ≥1 adverse event (AE) | Up to 24 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Percentage of participants with a Grade 3 or 4 AE | Up to 24 weeks
  Grade 3 or 4 AEs are "severe symptoms that cause inability to perform usual social and functional activities with intervention or hospitalization indicated (Grade 3), or "potentially life-threatenting events" (Grade 4).
Percentage of participants with overall mortality | Up to 24 weeks
  The percentage of participants with mortality through 24 weeks will be determined.
Percentage of participants discontinuing from study treatment due to an AE | Up to 24 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Percentage of participants discontinuing from study treatment due to a drug-related AE | Up to 24 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, that is considered to be related to DOR.

SECONDARY OUTCOMES:
Plasma concentration of DOR | Day 1 predose, Week 4 predose, Week 8 random, Week 12 random, and Week 24 predose and 0.5-2 hours postdose
  The DOR plasma concentration will be determined with sparse PK sampling.
Plasma concentration of 3TC | Day 1 predose, Week 4 predose, Week 8 random, Week 12 random, and Week 24 predose and 0.5-2 hours postdose
  The 3TC plasma concentration will be determined with sparse PK sampling.
Plasma concentration of TFV | Day 1 predose, Week 4 predose, Week 8 random, Week 12 random, and Week 24 predose and 0.5-2 hours postdose
  The TFV plasma concentration will be determined with sparse PK sampling.
AUC0-24hr of 3TC | Predose and 1, 2, 4, 12, and 24 hours postdose on Day 42
  Plasma AUC0-24 hr of 3TC will be determined at steady-state.
AUC0-24hr of TFV | Predose and 1, 2, 4, 12, and 24 hours postdose on Day 42
  Plasma AUC0-24 hr of TFV will be determined at steady-state.
Cmax of 3TC | Day 1 predose, Week 4 predose, Week 8 random, Week 12 random, and Week 24 predose and 0.5-2 hours postdose
  Plasma Cmax of 3TC will be determined.
Cmax of TFV | Day 1 predose, Week 4 predose, Week 8 random, Week 12 random, and Week 24 predose and 0.5-2 hours postdose
  Plasma Cmax of TFV will be determined.
Percentage of participants with ≥1 AE | Up to 48 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Percentage of participants with ≥1 AE | Up to 96 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Percentage of participants with Grade 3 or 4 AE | Up to 48 weeks
  Grade 3 or 4 AEs are "severe symptoms that cause inability to perform usual social and functional activities with intervention or hospitalization indicated (Grade 3), or "potentially life-threatenting events" (Grade 4).
Percentage of participants with Grade 3 or 4 AE | Up to 96 weeks
  Grade 3 or 4 AEs are "severe symptoms that cause inability to perform usual social and functional activities with intervention or hospitalization indicated (Grade 3), or "potentially life-threatenting events" (Grade 4).
Percentage of participants with overall mortality | Up to 48 weeks
  The percentage of participants with mortality through 48 weeks will be determined.
Percentage of participants with overall mortality | Up to 96 weeks
  The percentage of participants with mortality through 96 weeks will be determined.
Percentage of participants discontinuing from study treatment due to AE | Up to 48 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Percentage of participants discontinuing from study treatment due to AE | Up to 96 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Percentage of participants discontinuing from study treatment due to drug-related AE | Up to 48 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, that is considered to be related to DOR.
Percentage of participants discontinuing from study treatment due to drug-related AE | Up to 96 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, that is considered to be related to DOR.
Percentage of participants with human immunodeficiency virus type 1 (HIV-1) ribonucleic acid (RNA) <50 copies/mL | Up to 24 weeks
  Plasma HIV-1 RNA quantification will be performed at the central laboratory using a real-time polymerase chain reaction (PCR) assay with a lower limit of detection of 40 copies/mL.
Percentage of participants with HIV-1 RNA <50 copies/mL | Up to 48 weeks
  Plasma HIV-1 RNA quantification will be performed at the central laboratory using a real-time PCR assay with a lower limit of detection of 40 copies/mL.
Percentage of participants with HIV-1 RNA <50 copies/mL | Up to 96 weeks
  Plasma HIV-1 RNA quantification will be performed at the central laboratory using a real-time PCR assay with a lower limit of detection of 40 copies/mL.
Percentage of participants with HIV-1 RNA <200 copies/mL | Up to 24 weeks
  Plasma HIV-1 RNA quantification will be performed at the central laboratory using a real-time PCR assay with a lower limit of detection of 40 copies/mL.
Percentage of participants with HIV-1 RNA <200 copies/mL | Up to 48 weeks
  Plasma HIV-1 RNA quantification will be performed at the central laboratory using a real-time PCR assay with a lower limit of detection of 40 copies/mL.
Percentage of participants with HIV-1 RNA <200 copies/mL | Up to 96 weeks
  Plasma HIV-1 RNA quantification will be performed at the central laboratory using a real-time PCR assay with a lower limit of detection of 40 copies/mL.
Percentage of virologically-suppressed (VS) participants with HIV-1 RNA ≥50 copies/mL | Up to 24 weeks
  Plasma HIV-1 RNA quantification will be performed at the central laboratory using a real-time PCR assay with a lower limit of detection of 40 copies/mL.
Percentage of VS participants with HIV-1 RNA ≥50 copies/mL | Up to 48 weeks
  Plasma HIV-1 RNA quantification will be performed at the central laboratory using a real-time PCR assay with a lower limit of detection of 40 copies/mL.
Percentage of VS participants with HIV-1 RNA ≥50 copies/mL | Up to 96 weeks
  Plasma HIV-1 RNA quantification will be performed at the central laboratory using a real-time PCR assay with a lower limit of detection of 40 copies/mL.
Percentage of treatment-naive (TN) participants with log10 change from baseline in HIV-1 RNA | Day 1 and Week 24
  Plasma HIV-1 RNA quantification will be performed at the central laboratory using a real-time PCR assay with a lower limit of detection of 40 copies/mL.
Percentage of TN participants with log10 change from baseline in HIV-1 RNA | Day 1 and Week 48
  Plasma HIV-1 RNA quantification will be performed at the central laboratory using a real-time PCR assay with a lower limit of detection of 40 copies/mL.
Percentage of TN participants with log10 change from baseline in HIV-1 RNA | Day 1 and Week 96
  Plasma HIV-1 RNA quantification will be performed at the central laboratory using a real-time PCR assay with a lower limit of detection of 40 copies/mL.
Change from baseline in cluster of differentiation 4+ (CD4+) T-cell counts | Day 1 and Week 24
  Plasma HIV-1 RNA quantification will be performed at the central laboratory using a real-time PCR assay with a lower limit of detection of 40 copies/mL.
Change from baseline in CD4+ T-cell counts | Day 1 and Week 48
  Plasma HIV-1 RNA quantification will be performed at the central laboratory using a real-time PCR assay with a lower limit of detection of 40 copies/mL.
Change from baseline in CD4+ T-cell counts | Day 1 and Week 96
  Plasma HIV-1 RNA quantification will be performed at the central laboratory using a real-time PCR assay with a lower limit of detection of 40 copies/mL.
Viral resistance-associated substitutions (RASs) to DOR or other treatment components | Up to 96 weeks
  The presence of viral RASs to DOR or other treatment components will be monitored for up to 96 weeks.
Percentage of participants adhering to DOR treatment regimen | Up to 96 weeks
  Adherence to DOR will be monitored for up to 96 weeks.
Assessment of palatability/acceptability of DOR pellets/granules | Day 28
  Palatability/acceptability will be based on scores on the 5-point facial hedonic scale (FHS). FHS scores will be tabulated, and summarized by mean and SD, on Day 28. The highest possible FHS score is 5, with higher scores indicative of greater palatability.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (24):
- United States (2):
  - University of Colorado at Denver ( Site 0108), Aurora, Colorado
  - Emory Children's Center ( Site 0103), Atlanta, Georgia
- Colombia (3):
  - Clinica Somer ( Site 1003), Rionegro, Antioquia
  - Ciensalud Ips S A S ( Site 1001), Barranquilla, Atlántico
  - CEIP - Centro de Estudios en Infectología Pediátrica ( Site 1002), Cali, Valle del Cauca Department
- Mexico (3):
  - Hospital Infantil de Mexico Federico Gomez ( Site 0702), Mexico City, Mexico City
  - Unidad de Atencion Medica e Investigacion en Salud S.C. ( Site 0700), Mérida, Yucatán
  - Instituto Nacional de Pediatria ( Site 0701), Mexico City
- Russia (5):
  - Kuzbasskiy Center for the Prevention and Control of AIDS ( Site 0506), Kemerovo, Kemerovo Oblast
  - Clinical Centre for Prevention and Control of AIDS ( Site 0504), Krasnodar, Krasnodarskiy Kray
  - Krasnoyarsk Regional Center for Prevention and Control of AIDS ( Site 0507), Krasnoyarsk, Krasnoyarsk Krai
  - Infectious Clinical Hospital #2 ( Site 0501), Moscow, Moscow
  - FGU Republican Clinical Infectious Hospital of Roszdrav ( Site 0500), Saint Petersburg, Sankt-Peterburg
- South Africa (8):
  - FARMOVS PTY LTD ( Site 0601), Bloemfontein, Free State
  - Perinatal HIV Research Unit ( Site 0602), Johannesburg, Gauteng
  - Wits Reproductive Health and HIV Institute (WRHI) ( Site 0603), Johannesburg, Gauteng
  - Empilweni Services and Research Unit ( Site 0604), Johannesburg, Gauteng
  - King Edward Hospital ( Site 0600), Durban, KwaZulu-Natal
  - Family Clinic Research With UBUNTU ( Site 0605), Cape Town, Western Cape
  - Be Part Yoluntu Centre ( Site 0606), Paarl, Western Cape
  - Tsitsikamma Clinical Research Initiative (TCRI) ( Site 0607), Plettenberg Bay, Western Cape
- Thailand (3):
  - Siriraj Hospital ( Site 0901), Bangkok, Bangkok
  - Research Institute for Health Sciences ( Site 0902), Chiang Mai
  - Faculty of Medicine - Khon Kaen University ( Site 0903), Khon Kaen

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/